CLINICAL TRIAL: NCT06545539
Title: Does Participation in a Fall Preparedness Program Improve Fall Efficacy Among Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Collaborators: YMCA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-2
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Fall Injury; Fall; Falls (Accidents) in Old Age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fall Preparedness Class Participants (Experimental): Participants who meet inclusion and exclusion requirements of the study and sign an informed consent.
  Interventions: Other: Fall Preparedness Exercise Class

INTERVENTIONS:
Other: Fall Preparedness Exercise Class — The class will be held bi-weekly at two different locations. To ensure consistency across groups, the instructor(s) will adhere to a standardized class outline. Exercise modifications will be provided as necessary to adjust the intensity, ensuring all participants can follow the program.

SUMMARY:
The purpose of this study is to determine if a fall preparedness program can reduce the fear of falling in older adults and subsequently improve their function and reduce falls with injury.

Participants will perform baseline measures 4 weeks before intervention and again at the start of intervention. They will perform a 12-week intervention and then complete outcome measures again at the conclusion of the program.

DETAILED DESCRIPTION:
A. Methods and Procedures

1. Introduction Falls are a major concern with the growing older adult population in the US1. Falls lead to injury, reduced quality of life (QOL), fear of falling (FoF), institutionalization, morbidity, and mortality1. Many evidence-based programs exist to prevent falls, however the number of falls continues to rise1,2. There are no current programs that utilize the use of floor transfers and fall landing strategies to reduce the fear of falling in older adults.
2. Background

i. According to the CDC, falls are a leading cause of fatal and non-fatal injuries in older adults. Due to the increasing number of older adults, people aged sixty-five years or older, the number of falls is predicted to raise to 52 million per year by 20301. Falls cost the healthcare system $50 billion dollars annually, and that number is expected to rise with the growing number of older adults1. There are many causes that lead to falls, including weakness, vitamin D deficiency, osteoporosis, balance impairments, polypharmacy, vision impairments, foot deformities, foot pain, improper footwear, and hazards in home to name a few more common causes1. Falls can have many negative consequences, including brain injury, broken bones, and fear if falling1.

ii. Fear of falling (FoF) is described as a concern about falls that may lead to reduced balance confidence and reduced self-efficacy that can lead to limitations on daily activities2,3. FoF is present in 21-85% of the older adult population, in both fallers and non-fallers2. Reduced activity from the FoF can lead to a reduction in daily activities, that leads to weakness and reduced balance which can then cause a person to be a higher fall risk1. There is an increased risk for frailty in older adults who experience FoF4.

iii. Due to the vast list of causes of falls, there are many interventions available to treat falls and fall anxiety. Exercise interventions and programs such as tai chi, yoga, and the OTAGO have been described as mechanisms to reduce FoF2,5-7. Another option is a multifactorial program intervention that focuses on removal of trip hazards and medication review in addition to exercise7,8. Cognitive behavioral therapy and relaxation training may also be feasible treatments in reducing FoF in older adults9. A Matter of Balance is an evidenced based cognitive behavioral therapy program that helps reduce fear of falling10.

iv. One area that has not been thoroughly researched is the use of teaching safe fall landing strategies and the use of floor transfers to reduce their FoF as well as falls with injuries. A systematic review in 2017 by Moon and Sosnoff identified seven different strategies that were shown to reduce impact force during a fall11. These strategies include squatting, stepping, flexing elbows, forward rotation, martial arts rolling, and relaxing muscles11. Arkkukangas et al. implemented a Judo4Balance program, which incorporates martial arts falling techniques, and discovered that these techniques were effectively teachable to older adults12. Another study examined the use of martial arts falling techniques in older adults and found that these techniques significantly reduced the impact load on the hip and decreased the FoF13. The floor transfer test is a reliable measure to assess physical function and mobility in older adults and is an important piece of fall recovery training14,15. However, floor transfers are not always routinely taught to older adults by their various care providers14. It is unknown if education on floor transfers could improve fall efficacy in older adults.

c. Objectives The purpose of this study is to determine if a fall preparedness program can improve fall efficacy in older adults and subsequently increase activity level, reduce fall risk and falls with injury.

d. Study design and procedures i. How the participants will be identified and recruited and how informed consent will be obtained to minimize coercion or undue influence: The study design is a quasi-experimental, longitudinal cohort study. Older adults will be recruited through fliers posted throughout the community and online through social media, word of mouth, emails, and information on the affiliated website. All recruitment materials will provide clear, concise information about the study's purpose, procedures, risks, and benefits, and will emphasize that participation is entirely voluntary.

Interested participants will have the option to call the Department of Graduate Studies in Health and Rehabilitation Sciences or send an email to gain more information about the study. Student workers, who are not involved in the study, will be trained to provide unbiased information, answer questions, and accept registrations. This student worker will ensure that potential participants understand that their participation is voluntary and that they can withdraw at any time without penalty.

Once participants express interest, they will be provided with an informed consent document in person or through email that includes comprehensive details about the study. Participants will be encouraged to review the document at their own pace, discuss it with family or friends, and contact the research team with any questions before signing.

The informed consent process will repeatedly emphasize that participation is voluntary and that there are no negative consequences for choosing not to participate or for withdrawing from the study at any time. The process for expressing interest and registering for the study will maintain participant confidentiality, and no identifying information will be collected until participants have formally consented to join the study outside of phone numbers and email addresses.

ii. Procedures for data collection: Participants will be assessed 4 weeks before the study begins. During this initial assessment, we will collect demographic information, conduct the American College of Sports Medicine (ACSM) Preparticipation Screening Guidelines and vital assessment, record fall history, and gather scores for the Fall Efficacy Scale International (FES-I), Short Physical Performance Battery (SPPB), Physical Activity Scale for the Elderly (PASE), and the Six-Item Cognitive Impairment Test (6CIT). A licensed physical therapist will perform this assessment. All participants who meet the inclusion criteria will proceed to the second assessment and start the intervention.

The second assessment will occur at the start of the study, where we will collect FES-I, PASE, fall history, and SPPB scores again. A final assessment will be conducted after the intervention, using the same measures: FES-I, PASE, fall history, and SPPB.

Participants will be assigned a subject number during the initial data collection. There will be a link connecting the participants' name to their ID numbers on a master spreadsheet kept by the principal investigator on a password-protected university laptop computer. No identifying information will be included on any paper or computerized forms, only the participants' assigned ID number. All outcome testing will be conducted by a single investigator, who is a physical therapist.

During testing, participants will be asked if they are willing to participate in follow-up calls and interviews. Those who agree will be asked open-ended questions upon completing the intervention. These questions aim to explore their perspectives and emotions regarding fall efficacy, fear of falling, engagement in the intervention, and any perceived changes resulting from it. (The interview form is attached as Appendix A.) iii. Procedures to which human subjects will be exposed/ risks and benefits: Participants in this study will engage in exercise activities, which can induce various physiological changes, potentially leading to adverse reactions. These reactions may encompass injuries to muscles, tendons, ligaments, bones, and joints, as well as fluctuations in blood pressure, dizziness, fainting, and in exceedingly rare cases, cardiac rhythm disturbances, heart attacks, strokes, or even fatality. Every endeavor will be undertaken to mitigate these risks through thorough pre-exercise evaluations, continual supervision during exercises, and transparent communication regarding any discomfort or concerns experienced throughout the study.

Participation in this assessment and exercise class holds the potential to yield valuable data, which could be utilized to tailor an exercise regimen specifically suited to participant needs. Additionally, engagement in this program may foster a deeper comprehension of physical fitness and functional capacity, empowering participants with insights into personal physical boundaries and capabilities for engaging in physical activities.

iv. Intervention: The class will be held bi-weekly at two different locations, Youngstown State University in Youngstown, Ohio and the Davis Family YMCA in Boardman, Ohio. To ensure consistency across groups, the instructor(s) will adhere to a standardized class outline (Appendix C). Exercise modifications will be provided as necessary to adjust the intensity, ensuring all participants can follow the program.

v. Instructor: There will be one primary instructor and a substitute instructor. All instructors will either have a B.S. in exercise science or be licensed physical therapists. Instructors will be trained on the class expectations and format by Shannon Dudash (investigator). A detailed class format will be provided to the instructor (Appendix C). Outcome measure data will not be collected by the instructor but by a separate investigator.

vi. Data Analysis

1. Sample size and power: We conducted an a priori power analysis using G*Power with an effect size of 0.36 for a one-group F-test ANOVA, aiming for a power of 0.8, which resulted in a required sample size of 14. However, since the effect size was determined based solely on FES-I recommendations for older adults with and without cognitive impairments and considering the possibility of overestimating the effect in a single-group study, we have decided to increase the sample size to 3016.
2. Descriptive statistics will be used to calculate frequencies, means, standard deviations (SD), interquartile ranges (IQR), as well as minimum and maximum values to illustrate the central tendency of the data.
3. We plan to analyze data using repeated measures ANOVA for within-group differences across the three time points.

B. Human Research Participants I. Participants i. Inclusion criteria: Adults age 60 and up; able to participate in exercise program ii. Exclusion criteria: Adults age <60 year old, severe medical condition that prohibits the ability to participate in an exercise program; 6CIT score that indicates severely impaired cognition. Severe medical conditions will be screed by a licensed Physical Therapist. Under the Ohio Practice Act, physical therapists in Ohio are permitted to differently diagnosis. The class participants will be community-dwelling older adults who are less likely to come to participate in an exercise class if they have any severe medical conditions.

Any participants with mild cognitive impairment who are not excluded from the study will be offered simplified instructions by the licensed physical therapist performing the assessments. They will also be offered increased verbal, visual, and tactile cues as needed throughout the program to ensure understanding.

II. Recruitment Procedures

1. Convenience sampling will be used. Older adults will be recruited through fliers posted throughout the community, word of mouth, and online through social media, emails, and information on the affiliated website. Interested participants will call to register or gain more information about the study.
2. No coercion will be used in the recruitment process. C. Informed Consent and Assent

a. Informed consent is attached as Appendix B and to IRB application separately b. No minors, prisoners, or individuals with intellectual disabilities will be included in this study.

c. The record of informed consent will be stored in the primary contact's office in a locked filing cabinet.

D. Confidentiality of Information Collected

1. All outcome measures will be collected anonymously. No names of the participants will be collected except the informed consent form.
2. Data will be stored on a research laptop computer that is password protected. All signed informed consent forms will be stored in a locked file cabinet in a locked office on Youngstown State University Campus and will be shredded after 3 years in accordance with IRB standards.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 60 and up
* able to participate in exercise program

Exclusion criteria:

* Adults age <60 year old
* severe medical condition that prohibits the ability to participate in an exercise program
* 6CIT score that indicates severely impaired cognition.

Severe medical conditions will be screed by a licensed Physical Therapist. Under the Ohio Practice Act, physical therapists in Ohio are permitted to differently diagnosis. The class participants will be community-dwelling older adults who are less likely to come to participate in an exercise class if they have any severe medical conditions.

Any participants with mild cognitive impairment who are not excluded from the study will be offered simplified instructions by the licensed physical therapist performing the assessments. They will also be offered increased verbal, visual, and tactile cues as needed throughout the program to ensure understanding.

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fall Efficacy Scale International (FES-I) | 4 weeks before start of intervention through completion of intervention; approximately 15 weeks
  Measure of self reported fall efficacy

SECONDARY OUTCOMES:
short physical performance battery (SPPB) | 4 weeks before start of intervention through completion of intervention; approximately 15 weeks
  measure of physical performance
Physical Activity Scale for the Elderly (PASE) | 4 weeks before start of intervention through completion of intervention; approximately 15 weeks
  Measure of self reported activity level in older adults

OTHER OUTCOMES:
Six-item cognitive impairment test (6CIT) | 4 weeks before start of intervention
  cognitive impairment test used to rule out participants

CONTACTS AND LOCATIONS:
Overall Officials: Shannon J Dudash, Principal Investigator — Youngstown State University
Locations (2):
- United States (2):
  - YMCA, Boardman, Ohio
  - Youngstown State University, Youngstown, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feng C, Adebero T, DePaul VG, Vafaei A, Norman KE, Auais M. A Systematic Review and Meta-Analysis of Exercise Interventions and Use of Exercise Principles to Reduce Fear of Falling in Community-Dwelling Older Adults. Phys Ther. 2022 Jan 1;102(1):pzab236. doi: 10.1093/ptj/pzab236. PMID 34636923
- [Background] Liu M, Hou T, Li Y, Sun X, Szanton SL, Clemson L, Davidson PM. Fear of falling is as important as multiple previous falls in terms of limiting daily activities: a longitudinal study. BMC Geriatr. 2021 Jun 7;21(1):350. doi: 10.1186/s12877-021-02305-8. PMID 34098904
- [Background] de Souza LF, Canever JB, Moreira BS, Danielewicz AL, de Avelar NCP. Association Between Fear of Falling and Frailty in Community-Dwelling Older Adults: A Systematic Review. Clin Interv Aging. 2022 Feb 9;17:129-140. doi: 10.2147/CIA.S328423. eCollection 2022. PMID 35173427
- [Background] Kumar A, Delbaere K, Zijlstra GA, Carpenter H, Iliffe S, Masud T, Skelton D, Morris R, Kendrick D. Exercise for reducing fear of falling in older people living in the community: Cochrane systematic review and meta-analysis. Age Ageing. 2016 May;45(3):345-52. doi: 10.1093/ageing/afw036. PMID 27121683
- [Background] Schmid AA, Van Puymbroeck M, Koceja DM. Effect of a 12-week yoga intervention on fear of falling and balance in older adults: a pilot study. Arch Phys Med Rehabil. 2010 Apr;91(4):576-83. doi: 10.1016/j.apmr.2009.12.018. PMID 20382290
- [Background] Zijlstra GA, van Haastregt JC, van Rossum E, van Eijk JT, Yardley L, Kempen GI. Interventions to reduce fear of falling in community-living older people: a systematic review. J Am Geriatr Soc. 2007 Apr;55(4):603-15. doi: 10.1111/j.1532-5415.2007.01148.x. PMID 17397441
- [Background] Chua CHM, Jiang Y, Lim S, Wu VX, Wang W. Effectiveness of cognitive behaviour therapy-based multicomponent interventions on fear of falling among community-dwelling older adults: A systematic review and meta-analysis. J Adv Nurs. 2019 Dec;75(12):3299-3315. doi: 10.1111/jan.14150. Epub 2019 Aug 27. PMID 31287182
- [Background] Yoshikawa A, Ramirez G, Smith ML, Lee S, Ory MG. Systematic review and meta-analysis of fear of falling and fall-related efficacy in a widely disseminated community-based fall prevention program. Arch Gerontol Geriatr. 2020 Nov/Dec;91:104235. doi: 10.1016/j.archger.2020.104235. Epub 2020 Aug 18. PMID 32911232
- [Background] Moon Y, Sosnoff JJ. Safe Landing Strategies During a Fall: Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2017 Apr;98(4):783-794. doi: 10.1016/j.apmr.2016.08.460. Epub 2016 Aug 31. PMID 27592402
- [Background] Arkkukangas M, Stromqvist Baathe K, Ekholm A, Tonkonogi M. High Challenge Exercise and Learning Safe Landing Strategies among Community-Dwelling Older Adults: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Jun 16;19(12):7370. doi: 10.3390/ijerph19127370. PMID 35742618
- [Background] Groen BE, Smulders E, de Kam D, Duysens J, Weerdesteyn V. Martial arts fall training to prevent hip fractures in the elderly. Osteoporos Int. 2010 Feb;21(2):215-21. doi: 10.1007/s00198-009-0934-x. Epub 2009 May 1. PMID 19407919
- [Background] Swancutt DR, Hope SV, Kent BP, Robinson M, Goodwin VA. Knowledge, skills and attitudes of older people and staff about getting up from the floor following a fall: a qualitative investigation. BMC Geriatr. 2020 Oct 6;20(1):385. doi: 10.1186/s12877-020-01790-7. PMID 33023509
- [Background] Ardali G, Brody LT, States RA, Godwin EM. Reliability and Validity of the Floor Transfer Test as a Measure of Readiness for Independent Living Among Older Adults. J Geriatr Phys Ther. 2019 Jul/Sep;42(3):136-147. doi: 10.1519/JPT.0000000000000142. PMID 29059121
- [Background] Hauer KA, Kempen GI, Schwenk M, Yardley L, Beyer N, Todd C, Oster P, Zijlstra GA. Validity and sensitivity to change of the falls efficacy scales international to assess fear of falling in older adults with and without cognitive impairment. Gerontology. 2011;57(5):462-72. doi: 10.1159/000320054. Epub 2010 Oct 22. PMID 20975251
- See also: statistics and facts about falls in the older adult population — https://www.cdc.gov/falls/about/index.html